CLINICAL TRIAL: NCT03342014
Title: First Trimester Screening for Preeclampsia and Intrauterine Growth RestrIction Using Three Dimensional Doppler Angiography (SPIRIT): A Prospective Study in Nulliparous Pregnant Women
Brief Title: First Trimester Screening for Preeclampsia and Intrauterine Growth RestrIction Using Three Dimensional Doppler Angiography
Acronym: SPIRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Olivier MOREL, Professor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02418-45
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will have the same intervention (3DPD and UAD acquisitions ; blood sample)
  Interventions: Device: Ultrasound; Biological: Blood sample collection

INTERVENTIONS:
Device: Ultrasound — 3DPD and UAD acquisitions (10 min)
Biological: Blood sample collection — A blood sampling (20 mL) is collected for biomarker analysis (PAPP-A and PlGF) and biological collection.

SUMMARY:
Introduction: Preeclampsia (PE) and intrauterine growth restriction (IUGR) are two major pregnancy complications, related to a chronic utero-placental hypoperfusion. Nowadays, there isn't a screening or diagnostic test in clinic for utero-placental vascularization deficiency. Since 2004, 3D Power Doppler angiography has been used for the evaluation of utero-placental vascularisation and three vascular indices have been calculated: the vascularisation index (VI), flow index (FI) and vascularisation-FI (VFI). A high intra and inter-observer reproducibility and its potential interest for placental function study were reported. The investigator's main hypothesis is that these 3DPD indices could provide predictive values for PE and/or IUGR occurrence much higher than those observed with the currents other markers.

Objectives: The main objective of this study is to determine differences in 3DPD indices at first trimester between pregnancies defined at their outcome as uncomplicated pregnancy, PE (mild and severe) and IUGR in nulliparous women.

Methods and analysis: This is a prospective study. The investigators expect to include 2200 women in 4 French centers: Centre Hospitalier Universitaire de Nancy, Paris-Port-Royal (Assistance Publique - Hôpitaux de Paris), Strasbourg and Belfort (Hôpital Nord Franche-Comté).

The nulliparous pregnant women will be recruited during their 1st trimester consultation for routine Down syndrome screening (11-13+6 gestation weeks). Especially for the study, the 3DPD and Uterine Artery Doppler (UAD) acquisition, which last less than 10 min, will be included in the current routine 11-13+6 gestation weeks ultrasound screening. Also, additional blood samples will be taken for biomarker analysis (PAPP-A and P1GF) and biological collection. Utero-placental vascularization indices (VI, FI, VFI) will be quantified using VOCAL® software. For each subgroup (uncomplicated pregnancy, PE and IUGR) mean values in 3DPD indices will be computed and compared using a pairwise t test with a Bonferroni correction p value adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Singleton nulliparous pregnant women between 11 and 13+6 gestation weeks.
* Mandatory enrolment in a social security plan,
* Patient (or a third person, independent from the investigator and the sponsor, in case of inability to read or write) having signed an informed consent.

Exclusion Criteria:

* Patients under a measure of legal protection.
* Patient under 18,
* Absence of social insurance,
* Patient participating simultaneously to other interventional research trial to test a pharmaceutical treatment and protocols are not compatible,
* Inability to understand and accept the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2159 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Measure of 3D power Doppler indice : the vascularization index (VI) | through study completion, an average of 40 months
Measure of 3D power Doppler indice : the flow index (FI) | through study completion, an average of 40 months
Measure of 3D power Doppler indice : the vascularization-flow index (VFI) | through study completion, an average of 40 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertholdt C, Hossu G, Banasiak C, Beaumont M, Morel O. First trimester screening for pre-eclampsia and intrauterine growth restriction using three-dimensional Doppler angiography (SPIRIT): protocol for a multicentre prospective study in nulliparous pregnant women. BMJ Open. 2020 Oct 19;10(10):e037751. doi: 10.1136/bmjopen-2020-037751. PMID 33077562